CLINICAL TRIAL: NCT00092976
Title: A Phase IV Study of the Safety and Efficacy of ReFacto® (Moroctocog Alfa, B-Domain Deleted Recombinant Factor VIII) in Subjects With Hemophilia A Undergoing Major Surgery Monitored Using the Chromogenic Substrate Assay at the Local Laboratory
Brief Title: Study Evaluating ReFacto® in Hemophilia A Undergoing Major Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3082A2-401
Record Dates: First submitted 2004-09-28; First posted 2004-09-29 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2006-05

CONDITIONS: Hemophilia A
Keywords: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII SQ

INTERVENTIONS:
Drug: ReFacto

SUMMARY:
The primary objective of this clinical research study is to evaluate the safety and efficacy of ReFacto in subjects with hemophilia A undergoing major surgery monitored using the chromogenic substrate assay at the local laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 years
* Male previously treated patients (≥150 Exposure Days) with moderate or severe hemophilia A (i.e. ≤ 5% FVIII:C) who will undergo elective major surgery that is anticipated to require at least 6 consecutive days of daily factor VIII (FVIII) infusions (surgical and post-surgical prophylaxis)
* Ability to adhere to the protocol requirements

Exclusion Criteria:

* Hypersensitivity to ReFacto, murine allergen, or hamster allergen 2 History of FVIII inhibitor or current inhibitor, defined as > 0.6 BU
* Prior participation in this study
* Any concomitant bleeding disorder other than hemophilia A

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2003-02; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of ReFacto in subjects with Hemophilia A undergoing major surgery monitored using the chromogenic substrate assay at the local laboratory.

SECONDARY OUTCOMES:
To compare FVIII:C levels determined using the one-stage and the chromogenic substrate assays at a central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (4):
- United States (4):
  - Los Angeles, California
  - New Brunswick, New Jersey
  - Cincinnati, Ohio
  - Hershey, Pennsylvania